CLINICAL TRIAL: NCT04413786
Title: The Modulatory Effect of Oxytocin on Attentional Processing of Emotional Faces
Brief Title: Oxytocin's Effects on Face Attentional Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Shuxia Yao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-71
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: oxytocin; emotional faces; attention; N2pc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin group (Experimental): male subjects with oxytocin treatment
  Interventions: Drug: oxytocin treatment
- placebo group (Placebo Comparator): male subjects with placebo treatment
  Interventions: Drug: placebo treatment

INTERVENTIONS:
Drug: oxytocin treatment — intranasal administration of oxytocin (24IU)
  Arms: oxytocin group
Drug: placebo treatment — intranasal administration of placebo (24IU)
  Arms: placebo group

SUMMARY:
To investigate whether intranasal oxytocin (24IU) treatment has a regulatory effect on attentional processing of emotional faces.

DETAILED DESCRIPTION:
In a placebo-controlled double-blind between-subject design experiment, investigators plan to investigate the effect of oxytocin treatment on attentional processing of emotional faces. Subjects complete questionnaires in Chinese versions before treatment administration, including the Beck Depression Inventory, Autism Spectrum Quotient , Trait Anxiety Inventory, Toronto Alexithymia Scale, Multidimentional Assessment of Interoceptive Awareness. This experiment consists of two tasks including Emotional Face Cue-target Task and Visual Search Task. In the first task, subjects need to make a response to judge the position of target after a cue-target is presented. In the second task, subjects are asked to search the target "U" or inverted "U" placed on the nose of emotional/neutral faces and make an choices based on their oorientation. During these phases, subjects' response accuracy, response time and electrophysiological activity (ERP) are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders.

Exclusion Criteria:

* history of head injury
* medical or psychiatric illness

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-26 (Actual)

PRIMARY OUTCOMES:
Response time in reponse to different emotional face targets. | 1 hour
  Response time in discriminating which side (left or right) the emotional face target appear.
N2pc | 1 hour
  N2pc is an enhanced negative event-related potential typically elicited at posterior electrodes (e.g., PO7 and PO8) contralateral to the target presented among distractors between 180 and 300 ms after the onset of stimuli.
  display.

SECONDARY OUTCOMES:
Response accuracy in response to different emotional face targets. | 1 hour
  Response accuracy is caculated by the precentage of correct responses among the total responses in discriminating the position (left or right side) of different face conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Shuxia Yao, Doctor, Study Director — University of Electronic Science and Technology
Locations (1):
- School of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China